CLINICAL TRIAL: NCT01466361
Title: Evaluation of the Nicotine Lozenge in Relief of Provoked Acute Craving
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S7120994
Record Dates: First submitted 2011-11-03; First posted 2011-11-07 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Smoking; Smoking Cessation
Keywords: Nicotine; Nicotine craving
MeSH Terms: conditions — Smoking; Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lower dose Nicotine (Active Comparator): lower dose nicotine lozenge
  Interventions: Drug: Nicotine lower dose
- Higher dose Nicotine (Active Comparator): higher dose Nicotine lozenge
  Interventions: Drug: Nicotine higher dose
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotine lower dose — lower dose nicotine lozenge
  Arms: Lower dose Nicotine
Drug: Nicotine higher dose — higher dose nicotine lozenge
  Arms: Higher dose Nicotine
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
This study is designed to evaluate the ability of a nicotine lozenge to relieve craving for a cigarette compared to a matched placebo (a placebo is like sugar pill and contains no active).

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy smokers who smoke more than 5 cigarettes per day
* Body mass index (BMI) within the range 19-35 kilogram (kg)/meter (m)^2
* Females of childbearing potential who are, in the opinion of the investigator, practicing a reliable method of contraception.

Exclusion Criteria:

* Women who are pregnant or who have a positive urine pregnancy test.
* Participants with known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of their stated ingredients.
* Clinical Study/Experimental Medication: Participation in another clinical study or receipt of an investigational drug within 30 days of the screening visit.
* Prior Concomitant Medication: Treatment with enzyme altering agents (e.g. carbamazepine, phenytoin, cimetidine, sodium valporate) within 30 days of the craving provocation visit; Use of any prescription psychoactive medication (such as but not limited to antidepressants, antipsychotics, anxiolytics) within 14 days of the craving provocation visit; Participant has used an over-the-counter (OTC) medication such as antihistamines, sedating agents, or any compound that would have a sedating effect within 24 hours of the craving provocation visit; Current use of any nicotine replacement therapy.
* Substance abuse: Recent history or current history (within the last 1 year) of alcohol or other substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 187 (Actual)
Dates: Start 2010-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- Los Angeles Clinical Trials, Burbank, California, United States

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below)
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=19926

REFERENCES:
- [Derived] Nides M, Shanga GM, Bishop A, Becker WD. Nicotine Lozenges in the Relief of Behaviorally Provoked Craving. Am J Health Behav. 2018 May 1;42(3):69-80. doi: 10.5993/AJHB.42.3.7. PMID 29663982

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at the clinical site.
Pre-assignment Details: Participants who smoked more than 5 cigarettes per day were included in the study. Participants were stratified to treatments according to their smoking status: heavy smokers: smoking greater than 20 cigarettes per day and light smokers: smoking between 6 - 20 cigarettes per day.
Groups:
- Nicotine Lozenge 4 Milligrams (mg) (Heavy Smokers Group): Participants smoking more than 20 cigarettes per day, received a single dose of 4mg nicotine lozenge, through oral route.
- Placebo Lozenge (Heavy Smokers Group): Participants smoking more than 20 cigarettes per day, received a single dose of placebo lozenge, through oral route.
- Nicotine Lozenge 1.5mg (Light Smokers Group): Participants smoking between 6-20 cigarettes per day, received a single dose of 1.5mg nicotine lozenge, through oral route.
- Placebo Lozenge (Light Smokers Group): Participants smoking between 6-20 cigarettes per day, received a single dose of placebo lozenge, through oral route.
Period: Overall Study
Arm/Group | Nicotine Lozenge 4 Milligrams (mg) (Heavy Smokers Group) | Placebo Lozenge (Heavy Smokers Group) | Nicotine Lozenge 1.5mg (Light Smokers Group) | Placebo Lozenge (Light Smokers Group)
Started | 52 | 34 | 60 | 41
Completed | 52 | 34 | 60 | 41
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Nicotine Lozenge 4 mg (Heavy Smokers Group): Participants smoking more than 20 cigarettes per day, received a single dose of 4mg nicotine lozenge, through oral route.
- Placebo Lozenge 1 (Heavy Smokers Group): Participants smoking more than 20 cigarettes per day, received a single dose of placebo lozenge, through oral route.
- Placebo Lozenge 2 (Light Smokers Group): Participants smoking between 6-20 cigarettes per day, received a single dose of placebo lozenge, through oral route.
- Total: Total of all reporting groups
Arm/Group | Nicotine Lozenge 4 mg (Heavy Smokers Group) | Placebo Lozenge 1 (Heavy Smokers Group) | Nicotine Lozenge 1.5mg (Light Smokers Group) | Placebo Lozenge 2 (Light Smokers Group) | Total
Number analyzed (Participants) | 52 | 34 | 60 | 41 | 187
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.1 (10.42) | 45.9 (9.43) | 43.9 (11.48) | 45.0 (10.59) | 45.0 (10.48)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 16 | 24 | 21 | 84
  Male | 29 | 18 | 36 | 20 | 103
Nicotine cravings assessment baseline scores on a Visual Analogue scale (VAS) [Mean (Standard Deviation); unit: Score on a scale] — Participants were prohibited from smoking for 4 hours and then exposed to a provoked craving paradigm. During the provoked craving paradigm subjects were exposed to the sight and smell of a lit cigarette and were forbidden from putting the cigarette in their mouth. Cravings assessment was completed at the start of and immediately following the provoked craving paradigm using a VAS.
  Score on a scale
    Baseline score prior provoked craving paradigm(B1) | 68.3 (29.147) | 69.54 (26.534) | 70.00 (20.895) | 62.3 (25.785) | 67.5 (26.090)
    Baseline score post provoked craving paradigm (B2) | 76.03 (24.849) | 78.39 (23.659) | 76.96 (21.667) | 69.1 (26.335) | 75.1 (24.127)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Nicotine Cravings VAS Scores in Light Smokers
Description: Participants completed a nicotine craving assessment consisting of following five items: I have a desire for a cigarette right now, if it were possible I would smoke right now, All I want right now is a cigarette, I have an urge for a cigarette, I crave a cigarette right now. All participants indicated their craving intensity on a pre-drawn 100 mm scale ranging from 0 (disagree) to 100 (agree). At the end of the craving assessment period, mean VAS score (in mm) was measured.
Time Frame: Baseline, 1, 3, 5, 10 and 15 minutes post-treatment
Population: Intent to treat (ITT) population: All randomized participants with at least one cravings assessment measurement post dose were analyzed. No data was imputed in case of dropouts or missing data.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Nicotine Lozenge 1.5mg (Light Smokers Group): Participants smoking between 6-20 cigarettes/day, received a single dose of 1.5mg nicotine lozenge, through oral route.
- Placebo Lozenge 2 (Light Smokers Group): Participants smoking between 6-20 cigarettes/day, received a single dose of placebo lozenge, through oral route.
Arm/Group | Nicotine Lozenge 1.5mg (Light Smokers Group) | Placebo Lozenge 2 (Light Smokers Group)
Number analyzed (Participants) | 60 | 41
Score on a scale
  1 minute | -15.40 (2.439) | -8.17 (2.958)
  3 minutes | -24.42 (3.108) | -17.26 (3.770)
  5 minutes | -30.19 (3.257) | -23.86 (3.950)
  10 minutes | -35.33 (3.428) | -30.23 (4.158)
  15 minutes | -38.99 (3.689) | -33.99 (4.475)
Statistical Analysis 1: Comparison: Nicotine Lozenge 1.5mg (Light Smokers Group) vs Placebo Lozenge 2 (Light Smokers Group); Null hypothesis considered population means for treatments in comparison, to be equal with respect to provoked nicotine cravings at 1 minute post dosing; Test type: Superiority or Other; p = 0.0643, ANCOVA; Least square mean difference = -7.23, 95% CI 2-sided [-14.89 to 0.44] — Treatment comparisons were made between nicotine 1.5mg lozenge and placebo lozenge at 5% significance level
Statistical Analysis 2: Comparison: Nicotine Lozenge 1.5mg (Light Smokers Group) vs Placebo Lozenge 2 (Light Smokers Group); Null hypothesis considered population means for treatments in comparison, to be equal with respect to provoked nicotine cravings at 3 minute post dosing; Test type: Superiority or Other; p = 0.1489, ANCOVA; Least square mean difference = -7.16, 95% CI 2-sided [-16.93 to 2.61] — Treatment comparisons were made between nicotine 1.5mg lozenge and placebo lozenge at 5% significance level
Statistical Analysis 3: Comparison: Nicotine Lozenge 1.5mg (Light Smokers Group) vs Placebo Lozenge 2 (Light Smokers Group); Null hypothesis considered population means for treatments in comparison, to be equal with respect to provoked nicotine cravings at 5 minute post dosing; Test type: Superiority or Other; p = 0.2225, ANCOVA; Least square mean difference = -6.33, 95% CI 2-sided [-16.56 to 3.90] — Treatment comparisons were made between 1.5mg nicotine lozenge and placebo lozenge at 5% significance level
Statistical Analysis 4: Comparison: Nicotine Lozenge 1.5mg (Light Smokers Group) vs Placebo Lozenge 2 (Light Smokers Group); Null hypothesis considered population means for treatments in comparison, to be equal with respect to provoked nicotine cravings, 10 minutes post dosing; Test type: Superiority or Other; p = 0.3491, ANCOVA; Least square mean difference = -5.11, 95% CI 2-sided [-15.87 to 5.66] — Treatment comparisons were made between 1.5mg nicotine lozenge and placebo lozenge at 5% significance level
Statistical Analysis 5: Comparison: Nicotine Lozenge 1.5mg (Light Smokers Group) vs Placebo Lozenge 2 (Light Smokers Group); Null hypothesis considered population means for treatments in comparison, to be equal with respect to provoked nicotine cravings, 15 minutes post dosing; Test type: Superiority or Other; p = 0.3936, ANCOVA; Least square mean difference = -5.00, 95% CI 2-sided [-16.60 to 6.59] — Treatment comparisons were made between 1.5mg nicotine lozenge and placebo lozenge at 5% significance level

2. Primary Outcome: Mean Change From Baseline in Nicotine Cravings VAS Scores in Heavy Smokers
Description: as for outcome 1
Time Frame: Baseline, 3 minutes and 15 minutes post-treatment
Population: ITT population: All randomized participants who had at least one cravings assessment measurement post dose.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Groups:
- Nicotine Lozenge 4mg (Heavy Smokers Group): Participants smoking more than 20 cigarettes per day, received a single dose of 4mg nicotine lozenge, through oral route.
Arm/Group | Nicotine Lozenge 4mg (Heavy Smokers Group) | Placebo Lozenge 1 (Heavy Smokers Group)
Number analyzed (Participants) | 52 | 34
Score on a scale
  1 minute | -16.82 (2.613) | -13.24 (3.232)
  3 minutes | -29.52 (3.124) | -19.82 (3.865)
Statistical Analysis 1: Comparison: Nicotine Lozenge 4mg (Heavy Smokers Group) vs Placebo Lozenge 1 (Heavy Smokers Group); Null hypothesis considered population means for treatments in comparison, to be equal with respect to provoked nicotine cravings, at 1 minute post dosing; Test type: Superiority or Other; p = 0.3922, ANCOVA; Least square mean difference = -3.58, 95% CI 2-sided [-11.85 to 4.70] — Treatment comparisons were made between 4mg nicotine lozenge and placebo lozenge at 5% significance level
Statistical Analysis 2: Comparison: Nicotine Lozenge 4mg (Heavy Smokers Group) vs Placebo Lozenge 1 (Heavy Smokers Group); Null hypothesis considered population means for treatments in comparison, to be equal with respect to provoked nicotine cravings, 3 minutes post dosing; Test type: Superiority or Other; p = 0.0547, ANCOVA; Least square mean difference = -9.70, 95% CI 2-sided [-19.59 to 0.20] — Treatment comparisons were made between 4mg nicotine lozenge and placebo lozenge at 5% significance level

3. Secondary Outcome: Percentage of Responders With Improved Craving Scores in Heavy and Light Smokers Group
Description: Responders were defined as participants with an increase of at least one point (on the 100 point VAS scale) from baseline prior to provoked craving paradigm (B1) to baseline post provoked craving paradigm (B2) on the average cravings score. Percentage of these responders was calculated to evaluate the provocation rate.
Time Frame: Baseline prior to provoked craving paradigm, baseline post provoked craving paradigm
Measure: Number; unit: percentage
Groups:
- Light Smokers Group: Participants smoking between 6-20 cigarettes per day at baseline and responded to nicotine craving provocative paradigm before treatment
- Heavy Smokers Group: Participants smoking more than 20 cigarettes per day at baseline and responded to nicotine craving provocative paradigm before treatment
Arm/Group | Light Smokers Group | Heavy Smokers Group
Number analyzed (Participants) | 101 | 86
percentage | 77.2 | 75.6

4. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious AEs (SAEs)
Description: AE was defined as any new untoward medical occurrence or worsening of a pre-existing medical condition which does not necessarily have a causal relationship with study treatment/s.
  SAE was defined as any untoward medical occurrence that at any dose results in death; is life threatening; requires hospitalization or prolongation of existing hospitalization results in disability/ incapacity; is a congenital anomaly/ birth defect.
Time Frame: Baseline, 0 minute, 60 minutes and 5 days post treatment
Population: Safety population: All randomized participants who received the study treatments were considered evaluable for safety.
Measure: Number; unit: participants
Arm/Group | Nicotine Lozenge 4 mg (Heavy Smokers Group) | Placebo Lozenge 1 (Heavy Smokers Group) | Nicotine Lozenge 1.5mg (Light Smokers Group) | Placebo Lozenge 2 (Light Smokers Group)
Number analyzed (Participants) | 52 | 34 | 60 | 41
participants
  AEs | 11 | 0 | 1 | 1
  SAE | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: All AEs encountered or spontaneously reported following administration of any study treatment, and up to 5 days after the last administration of study treatment were recorded.
Arm/Group | Nicotine Lozenge 1.5mg (Light Smokers Group) | Nicotine Lozenge 4mg (Heavy Smokers Group) | Placebo Lozenge 1 (Heavy Smokers Group) | Placebo Lozenge 2 (Light Smokers Group)
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/52 | 0/34 | 0/41
Other Adverse Events (participants affected / at risk) | 1/60 | 11/52 | 0/34 | 1/41
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Lozenge 1.5mg (Light Smokers Group) (N=60) | Nicotine Lozenge 4mg (Heavy Smokers Group) (N=52) | Placebo Lozenge 1 (Heavy Smokers Group) (N=34) | Placebo Lozenge 2 (Light Smokers Group) (N=41)
Nausea (Gastrointestinal disorders) | 0 (0) | 5 (7) | 0 (0) | 0 (0)
Oral discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Throat Irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.